CLINICAL TRIAL: NCT05007028
Title: Nitrous Oxide for Late-Life Depression : a Randomized Controlled Trial With Comparator - PROTO-BRAIN
Brief Title: Nitrous Oxide for Late-Life Depression - PROTO-BRAIN
Acronym: PROTO-BRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR180133; 2019-002769-37 (EudraCT Number)
Record Dates: First submitted 2021-05-27; First posted 2021-08-16 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Late-Life Depression; Resistant Depression, Treatment
Keywords: Nitrous Oxide; Magnetic Resonance Imaging; Ultrasound Tissue Pulsatility Imaging
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Air

STUDY DESIGN:
Intervention Model Description: Randomized double blind trial with comparator
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrous Oxide (Experimental): Active Drug: EMONO (Equimolar Mixture of Oxygen and Nitrous Oxide)
  Interventions: Drug: EMONO
- Medical air (Placebo Comparator): Control Drug: Medical air : 78% N2 / 22% O2
  Interventions: Drug: Medical Air

INTERVENTIONS:
Drug: EMONO — Exposure to 1 hour of EMONO via facial mask
  Arms: Nitrous Oxide
Drug: Medical Air — Exposure to 1 hour of Medical Air via facial mask
  Arms: Medical air

SUMMARY:
Resistant Depression is a common condition in older adults and there is an urgent need for novel antidepressant in this population. Nitrous Oxide (N2O) has recently shown rapid antidepressant effect in midlife depression but no study has currently investigated the efficacy and safety of N2O in Late-Life Depression (LLD), while N2O may prove to be an ideal treatment for LLD because of glutamatergic antagonism and cerebrovascular effects and also a relatively good safety profile.

The goal of our study is to compare changes in depressive symptoms after 2 hours, 24 hours, 1 week and 2 week of a 1-hour exposure to EMONO (Equimolar Mixture of Oxygen and Nitrous Oxide) versus Medical Air.

Secondary Objectives include comparing differences in neuroimaging measures between 3 groups (responders and non-responders in the EMONO group, and patients in the control group).

DETAILED DESCRIPTION:
Secondary objectives include:

* To compare changes in Brain Tissue Pulsatility (BTP) as measured with Ultrasound Tissue Pulsatility Imaging (TPI) between responders in the EMONO group (MADRS change of at least 50%), non-responders in the EMONO group (MADRS change of no more than 50%) and in the Air Medical group
* To compare baseline differences in structural (brain volumes, white matter hyperintensities) and functional (resting state connectivity in BOLD, Brain Pulsatility in BOLD, Brain Perfusion in ASL) among the 3 groups
* To compare changes in depressive and anxiety symptoms between the active and control group, as assess with Hamilton scale, CGI scale, QIDS-SR, VAS and the STAI scale
* To compare safety between the active and control group, as assessed with SSI, YMRS, CADSS, BPRS

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-90 years-old
* Major Depressive Episode according to DSM-5 criteria, confirmed by the MINI - Mini International Neuropsychiatric Interview
* MADRS score greater than 20 (Montgomery Asberg Depression Rating Scale)
* Patient resistant to at least one well-conducted antidepressant treatment, as documented by the MGH-ATRQ scale
* Patient who can undergo N2O diffusion via a facial mask
* Patient who has signed an informed consent
* Person affiliated with a social security scheme

Exclusion Criteria:

* Bipolar disorder, schizophrenic disorder, neurodegenerative disease, documented by the MINI and the MMSE (non-inclusion if MMSE < 24/30), addictive disorder
* Unstable somatic pathology (including unstable neurological or cardiological diseases at risk of interfering with N2O diffusion)
* Presence of active and significant psychotic symptoms, at investigator's discretion
* Contraindications to EMONO (50%N2O/ 50%O2) : pneumothorax, emphysema, bowel obstruction, intracranial hypertension, chronic deficiency in vitamin B12 or B9
* Contraindications to MRI, including claustrophobia
* Legal incapacity and/or other circumstances unabling the patient to understand the nature, purpose or consequences of the study
* A person participating in a drug clinical trial or during a period of exclusion from any clinical study

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Change in MADRS | Baseline, 2 hours, 24 hours, 1 week, 2 weeks
  montgomery asberg depression scale for symptoms severity

SECONDARY OUTCOMES:
Change in Brain Tissue Pulsatility | Baseline and immediately after the intervention
  Indexes of BTP, including BTP amplitudes
MRI | At Baseline
  Structural and Functional MRI
Change in HDRS 17 items | Baseline, 2 hours, 24 hours, 1 week, 2 weeks
  Hamilton Depression Rating Scale
Change in QIDS-SR | Baseline, 2 hours, 24 hours, 1 week, 2 weeks
  Quick Inventory of Depressive Symptomatology Self Report, Depression severity
Change in CGI | Baseline, 2 hours, 24 hours, 1 week, 2 weeks
  Clinical Global Impression
Change in VAS | Baseline, 2 hours, 24 hours, 1 week, 2 weeks
  Visual Analog Scale for global well-being self assessement
Change in STAI | Baseline, 2 hours, 24 hours, 1 week, 2 weeks
  State-Trait Anxiety Inventory
Change in SSI | Baseline, 2 hours, 24 hours, 1 week, 2 weeks
  Scale for Suicidal Ideation
Change in YMRS | Baseline, 2 hours, 24 hours, 1 week, 2 weeks
  Young Mania Rating Scale
Change in Clinician Administered Dissociative States Scale | Baseline, 2 hours, 24 hours, 1 week, 2 weeks
  CADSS
Change in BPRS | Baseline, 2 hours, 24 hours, 1 week, 2 weeks
  Brief Psychiatric Rating Scale

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Tours, Tours, France